CLINICAL TRIAL: NCT00003505
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Primary Central Nervous System Lymphoma
Brief Title: Antineoplaston Therapy in Treating Patients With Primary Central Nervous System Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-LY-12; CDR0000066545 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-10

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — antineoplaston A10; antineoplaston AS 2-1; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally-occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating patients with primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety and possible effectiveness of antineoplastons A10 and AS2-1 in patients with serious or immediately life-threatening primary central nervous system lymphoma.
* Describe response to, tolerance to, and side effects of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gradually escalating doses of intravenous antineoplaston A10 and antineoplaston AS2-1 6 times per day until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with responding or stable disease may continue treatment.

Tumors are measured every 2 months for 6 months, every 3 months for 2 years, every 6 months for years 3 and 4, and then annually for years 5 and 6.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-IV primary central nervous system lymphoma for which no curative therapy exists
* Measurable tumor by MRI or CT scan
* Tumor must be greater than 2 cm in largest diameter

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2,000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic insufficiency

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No cardiac insufficiency
* No hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 4 weeks after study participation
* No serious infection requiring antibiotics, antifungals, or antivirals

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agents (e.g., interferon or interleukin-2)

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agent

Endocrine therapy:

* Concurrent corticosteroids allowed
* Must be on stable dose for at least 4 weeks prior to study entry

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplastons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States